CLINICAL TRIAL: NCT05951244
Title: Cathodal Transcranial Direct Current Stimulation in Patients With Drug-resistant Focal Epilepsy: Randomized Controlled Clinical Trial
Brief Title: Cathodal Transcranial Direct Current Stimulation in Patients With Drug-resistant Focal Epilepsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Koç University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NM002
Record Dates: First submitted 2023-03-30; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-04

CONDITIONS: Drug Resistant Epilepsy
Keywords: drug resistant epilepsy; transcranial direct current stimulation (tDCS)
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transcranial Direct Stimulation (Active Comparator): 20 epilepsy patients who were eligible and gave consent according to the inclusion criteria. For active group, tDCS treatment will be 2 mA current strength for 30 minutes.
  Interventions: Device: Transcranial Direct Current Stimulation-TessaNova (Teknofil-Turkiye)
- Sham-Transcranial Direct Current Stimulation (Sham Comparator): 20 epilepsy patients who were eligible and gave consent according to the inclusion criteria.
  For the sham group, the current will increase to 2mA in 10 seconds, continue for the 30s, then decrease to 0 in 10 seconds and cut off.
  Interventions: Device: Transcranial Direct Current Stimulation-TessaNova (Teknofil-Turkiye)

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation-TessaNova (Teknofil-Turkiye) — Sponge electrodes 5 x 7 cm in size will be used for tDCS application. The sponge electrodes will be wetted with saline and the cathode electrode will be placed on the seizure focus determined by EEG recording and seizure clinic, while the anode electrode will be placed on the contralateral shoulder-deltoid muscle.

SUMMARY:
The basis of this project is the application of cathodal tDCS in patients with drug-resistant focal epilepsy including patients whose seizures persist after epilepsy surgery, who rejected epilepsy surgery, and/or who are not suitable for surgery. For this purpose, 5-day consecutive cathodal electrical stimulation sessions will be used with personalized electrode montage according to the patient's seizure focus. In this context, the changes in seizures frequency and epileptic discharges will be examined for the first week and 12th week after the tDCS sessions through the seizure diary of the patients and the electroencephalogram (EEG) recordings to be taken. In addition, changes in cognitive functions, mood, and quality of life will be examined in patients after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older,
* Diagnosed with focal epilepsy with epileptic focus determined according to clinical and electroencephalogram recordings, who have undergone epilepsy surgery but seizures persist, who refuse epilepsy surgery or who are considered unsuitable for surgery,
* Patients who comply with the definition of drug-resistant epilepsy according to ILAE (International League Against Epilepsy Classification) criteria (Patients who have failed to achieve long-term seizure-free status despite at least two appropriate antiepileptic drugs given alone or in combination),
* Minimum 1 or more seizures per month (minimum 3 months),
* No antiepileptic dose change until 3 weeks before the study, stable treatment, and no dose change planned during the study,
* At least 1.5 Tesla MR imaging was performed before the study,
* Signed the informed consent form or the consent form signed by the legal representative,
* EEG was present before the study and all EEG data was accessible,
* Cooperative patients who can speak, understand and communicate in Turkish will be recruited.

Exclusion Criteria:

* The presence of any disease/deformity in the patient that the researchers believe will affect the patient's safety or the reliability of the data to be collected,
* Detection of more than one seizure focus in the patient,
* The patient had a psychogenic non-epileptic seizure attack (Psychogenic Non-epileptic Seizures -PNES) within 2 years prior to the study,
* Having a generalized onset seizure,
* Having had status epilepticus in the last 1 year,
* Presence of any disease, medical condition, or physical condition that, according to the researchers, could prevent, limit, affect or reduce the subject's completion of a minimum period of 1 + 12 weeks,
* Tissue damage (eczema, etc.) in the area where tDCS will be applied on the skin,
* Patients who are pregnant and do not use/do not want to use contraception during the study period,
* Lactating women,
* Metal implants, fillings in the head or teeth, presence of a medical device in the body (pacemaker, deep brain stimulator, cochlear implant, nerve stimulator, etc.)
* Presence of a skull defect with a radius of 5 mm and/or larger remaining from previous surgeries,
* The patient is participating in another clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Changes in epileptic discharge frequency at 1st week after tDCS compared to baseline epileptic discharge frequency | At the 1st week of follow-up after tDCS
  EEG recordings will be obtained after tDCS sessions. Epileptic discharges will be calculated from 30 minutes recordings. EEG will be recorded with scalp electrodes using a 128-channel Natus Quantum (Natus Medical) with a sampling rate 2048 Hz and 21 channels.
Changes in epileptic discharge frequency at 12th week after tDCS compared to baseline epileptic discharge frequency | At the 12th week of follow-up after tDCS
  EEG recordings will be obtained after tDCS sessions. Epileptic discharges will be calculated from 30 minutes recordings. EEG will be recorded with scalp electrodes using a 128-channel Natus Quantum (Natus Medical) with a sampling rate 2048 Hz and 21 channels.
Changes in epileptic seizure frequency at 12th week after tDCS compared to baseline (before the tDCS) | 3 months follow-up after tDCS
  The seizure diary of the patients will be recorded for 3 months follow-up after tDCS sessions. The seizure frequency will be evaluated in comparison to pre-tDCS seizure frequency.

SECONDARY OUTCOMES:
Quality of Life in Epilepsy Inventory (QOLIE-31) | At the 1st week and 12th week of follow-up after tDCS
  The QOLIE-31 is used to measure quality of life in epilepsy. The scale is scored between 0-100. A high score reflects a high quality of life.
Depression Anxiety and Stress Scale 21 (DASS-21) | At the 1st week and 12th week of follow-up after tDCS
  The DASS-21 is a self-report scale designed to measure the negative emotional states of depression, anxiety and stress. Individuals read each statement and circle a number 0, 1, 2 or 3 that indicates how much the statement is expressing his/her emotional state over the past week. The scale includes 21 questions and measure depression, stress and anxiety dimensions. A high score on the DASS- 21 indicates an increase in depression, anxiety and stress symptoms.
Pittsburgh Sleep Quality Index (PSQI) | At the 1st week and 12th week of follow-up after tDCS
  The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances. Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by summing the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.
Epworth Sleepiness Scale | At the 1st week and 12th week of follow-up after tDCS
  The Epworth Sleepiness Scale can be used to assess daytime sleepiness. It consists of a total of 8 questions. Each question is self-assessed by the patient with a number from 0 to 3. Scores can be interpreted as follows: 0-5 lower normal daytime sleepiness. 6-10 normal daytime sleepiness. 11-12 mild excessive daytime symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Ezgi Tuna Erdoğan, Assist Prof., Principal Investigator — Koç University School of Medicine
Locations (1):
- Koc University, Istanbul, Sarıyer, Turkey (Türkiye)